CLINICAL TRIAL: NCT06201312
Title: Effects of Crossover Point Exercise on Vascular Function of Women in Different Menopausal Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EOCPEOVFOWIDMY
Record Dates: First submitted 2023-12-07; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Vascular Health
Keywords: vascular health; crossover point

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early Postmenopausal Exercise Group (EE) (Experimental)
  Interventions: Other: COP exercise
- Late Postmenopausal Exercise Group (LE) (Experimental)
  Interventions: Other: COP exercise
- Early Postmenopausal Control Group (EC) (No Intervention)
- Late Postmenopausal Control Group (LC) (No Intervention)

INTERVENTIONS:
Other: COP exercise — crossover point intensity exercise
  Arms: Early Postmenopausal Exercise Group (EE); Late Postmenopausal Exercise Group (LE)

SUMMARY:
Recruit postmenopausal women and randomly assign them to one of four groups: Early Postmenopausal Exercise Group (EE), Late Postmenopausal Exercise Group (LE), Early Postmenopausal Control Group (EC), and Late Postmenopausal Control Group (LC).

All participates will undergo a graded exercise test to determine their maximum oxygen uptake, and vascular function response will be measured immediately after the exercise test. The COP exercise intensity for postmenopausal women will be obtained through the exercise test, and subjects in the EE and LE groups will undergo exercise training at this intensity for a period of three months. Tests and analyses of relevant indicators will be conducted on subjects in all four groups before and after the intervention. The exercise load experiments will be performed on a cycle ergometer.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women without cardiovascular disease

Exclusion Criteria:

* Women with undetermined menopause
* BMI <18.5 kg/m2 or BMI >28 kg/m2
* fasting plasma triglyceride levels ≥500 mgdl
* diabetes mellitus or fasting glucose >140 mgd
* blood creatinine >2.0 mgdl
* uncontrolled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >110 mmHg)
* untreated thyroid disease
* life-threatening illness with a prognosis of <5 years;
* history of deep vein thrombosis,
* pulmonary embolism, or breast cancer;
* currently receiving estrogen therapy.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Brachial Artery Flow-Mediated Dilation | 12 weeks
  The changes in brachial artery flow-mediated dilation are assessed at three time points: before the intervention, after the acute exercise, and three months following the intervention.
Carotid Intima-Media Thickness | 12 weeks
  The change of Carotid Intima-Media Thickness before and after intervention.
Carotid Diameter | 12 weeks
  The change of Carotid Diameter before and after intervention.
Carotid End-Diastolic Velocity | 12 weeks
  The change of Carotid End-Diastolic Velocity before and after intervention.
Carotid Peak Systolic Velocity | 12 weeks
  The change of Carotid Peak Systolic Velocity before and after intervention.
Pulsatility Index | 12 weeks
  The change of Pulsatility Index before and after intervention.
Resistive Index | 12 weeks
  The change of Resistive Index before and after intervention
Brachial-Ankle Pulse Wave Velocity | 12 weeks
  The change of Brachial-Ankle Pulse Wave Velocity before and after intervention.
Ankle-Brachial Index | 12 weeks
  The change of Ankle-Brachial Index before and after intervention.

SECONDARY OUTCOMES:
Serum Nitric Oxide level | 12 weeks
  The change of serum nitric oxide before and after intervention.
Plasma Nitrate level | 12 weeks
  The change of plasma nitrate before and after intervention.
ERRα mRNA and Protein Expression level | 12 weeks
  The change of ERRα mRNA and Protein Expression before and after intervention.
PGC1α mRNA Expression level | 12 weeks
  The change of PGC1α mRNA Expression before and after intervention
PGC1α Protein Expression level | 12 weeks
  The change of PGC1α Protein Expression before and after intervention
ERα mRNA Expression level | 12 weeks
  The change of ERα mRNA Expression before and after intervention
ERα Protein Expression level | 12 weeks
  The change of Protein Expression before and after intervention
p38MAPK mRNA Expression level | 12 weeks
  The change of p38MAPK mRNA Expression before and after intervention
p38MAPK Protein Expression level | 12 weeks
  The change of p38MAPK Protein Expression before and after intervention
Serum Reduced Glutathione level | 12 weeks
  The change of Serum Reduced Glutathione before and after intervention
Oxidized Glutathione level | 12 weeks
  The change of Oxidized Glutathione before and after intervention
Calculate GSSG/GSH Ratio | 12 weeks
  The change of Calculate GSSG/GSH Ratio before and after intervention
Serum Soluble Vascular Cell Adhesion Molecule-1 level | 12 weeks
  The change of Serum Soluble Vascular Cell Adhesion Molecule-1 Expression before and after intervention
Soluble Intercellular Adhesion Molecule-1 level | 12 weeks
  The change of Soluble Intercellular Adhesion Molecule-1 before and after intervention
Vascular Endothelial Growth Factor level | 12 weeks
  The change of Vascular Endothelial Growth Factor before and after intervention
body weight | 12 weeks
  The change of body weight before and after intervention
body mass index | 12 weeks
  The change of body mass index before and after intervention
Total Cholesterol level | 12 weeks
  The change of Total Cholesterol before and after intervention
Triglycerides level | 12 weeks
  The change of Triglycerides before and after intervention
High-Density Lipoprotein Cholesterol level | 12 weeks
  The change of High-Density Lipoprotein Cholesterol before and after intervention
Low-Density Lipoprotein Cholesterol level | 12 weeks
  The change of Low-Density Lipoprotein Cholesterol before and after intervention
Apolipoprotein AI level | 12 weeks
  The change of Apolipoprotein AI before and after intervention
Apolipoprotein B level | 12 weeks
  The change of Apolipoprotein B before and after intervention
Lipoprotein(a) level | 12 weeks
  The change of Lipoprotein(a) before and after intervention
Interleukin 6 level | 12 weeks
  The change of Interleukin 6 before and after intervention
Estradiol level | 12 weeks
  The change of Estradiol before and after intervention
Interventricular Septum Thickness in Systole | 12 weeks
  The change of Interventricular Septum Thickness in Systole before and after intervention
Interventricular Septum Thickness in Diastole | 12 weeks
  The change of Interventricular Septum Thickness in Diastole before and after intervention
Left Ventricular End-Systolic Diameter | 12 weeks
  The change of Left Ventricular End-Systolic Diameter before and after intervention
Left Ventricular End-Diastolic Diameter | 12 weeks
  The change of Left Ventricular End-Diastolic Diameter before and after intervention
Left Ventricular Posterior Wall Thickness in Systole | 12 weeks
  The change of Left Ventricular Posterior Wall Thickness in Systole before and after intervention
Left Ventricular Posterior Wall Thickness in Diastole | 12 weeks
  The change of Left Ventricular Posterior Wall Thickness in Diastole before and after intervention
Left Ventricular End-Systolic Volume | 12 weeks
  The change of Left Ventricular End-Systolic Volume before and after intervention
Left Ventricular End-Diastolic Volume | 12 weeks
  The change of Left Ventricular End-Diastolic Volume before and after intervention
Fractional Shortening | 12 weeks
  The change of Fractional Shortening before and after intervention
Left Ventricular Ejection Fraction | 12 weeks
  The change of Left Ventricular Ejection Fraction before and after intervention
Stroke Volume | 12 weeks
  The change of Stroke Volume before and after intervention
Heart Rate | 12 weeks
  The change of Heart Rate before and after intervention
Early Diastolic Mitral Inflow Velocity | 12 weeks
  The change of Early Diastolic Mitral Inflow Velocity before and after intervention
Atrial Diastolic Mitral Inflow Velocity | 12 weeks
  The change of Atrial Diastolic Mitral Inflow Velocity before and after intervention
Ratio of Early to Atrial Diastolic Mitral Inflow Velocity | 12 weeks
  The change of Ratio of Early to Atrial Diastolic Mitral Inflow Velocity before and after intervention
Cardiac Output | 12 weeks
  The change of Cardiac Output before and after intervention
NT-proBNP level | 12 weeks
  The change of NT-proBNP before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, China